CLINICAL TRIAL: NCT02908919
Title: Impact of Time Intervals on Quality and Tolerance of the Bowel Preparation
Brief Title: Impact of Time Intervals of Preparation on Quality and Tolerance of the Bowel Preparation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Collaborators: Nemocnice T.Bati, Zlin (Unknown); Brno University Hospital (Other); University Hospital, Motol (Other)
Responsible Party: Principal Investigator, MUDr. Jan Matous, Jan Matous, MD, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CB1601
Record Dates: First submitted 2016-09-09; First posted 2016-09-21 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Bowel Preparation; Colonoscopy
Keywords: Colonoscopy; Picosulfate sodium; Polyethylene glycol; Magnesium citrate; Ascorbic acid; SPMC (solution picosulfate + magnesium citrate); PEGA (Polyethylene glycol + ascorbic acid)
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fortrans pulv. sol (Active Comparator): Polyethylene glycol solution. Used 4 l before colonoscopy. Bowel preparation interval: QD/BID or one day.
  Interventions: Procedure: Colonoscopy
- Picoprep pulv. sol. (Active Comparator): Natrium picosulfate/ magnesium citrate solution. Used 2 l before colonoscopy. bowel preparation interval: QD/BID or one day.
  Interventions: Procedure: Colonoscopy
- Moviprep pulv. sol. (Active Comparator): Polyethylene glycol + ascorbic acid solution. Used 2 l before colonoscopy. Bowel preparation interval: QD/BID or one day.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — The quality of bowel preparation, which is checked during colonoscopy

SUMMARY:
The purpose of this study is to determine optimal time intervals for preparation before colonoscopy using different formulas.

DETAILED DESCRIPTION:
Different formulas are used for bowel preparation before colonoscopy. Present guidelines are based on conventional polyethylene glycol. Their validity for other preparations were not evaluated. Relationship between length of preparation, interval to colonoscopy and bowel preparation quality, tolerance are assessed.

ELIGIBILITY:
Inclusion Criteria:

- subjects referred to diagnostic or therapeutic colonoscopy.

Exclusion Criteria:

* ileus
* known or suspected bowel obstruction
* active bowel inflammation
* pregnancy
* any presence of serious medical conditions ( esp. cardiac, renal, liver diseases)
* history of prior colonic or rectal surgery
* inability to obtain valid data from

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of bowel preparation according to time intervals of bowel preparation | One day
  The length of bowel preparation and interval to colonoscopy for bowel preparation quality Aronchick score excellent and good

SECONDARY OUTCOMES:
Tolerance of bowel preparation according to time intervals of bowel preparation | One day

CONTACTS AND LOCATIONS:
Overall Officials: Jan Matous, MD, Principal Investigator — Faculty Hospital Kralovske Vinohrady, Prague
Locations (2):
- Czechia (2):
  - Faculty Hospital Kralovske Vinohrady, Prague
  - Nemocnice T.Bati, Zlín

IPD SHARING:
Plan to Share IPD: No